CLINICAL TRIAL: NCT06524544
Title: A Phase III Randomized Trial of Pembrolizumab in Combination With Sacituzumab Govitecan vs Standard of Care in Anti-PD(L)1-Resistant Advanced Urothelial Cancer
Brief Title: A Study Comparing the Combination of Pembrolizumab and Sacituzumab Govitecan Versus Standard of Care in the Treatment of Advanced Urothelial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-06208; NCI-2024-06208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8231 (Other: ECOG-ACRIN Cancer Research Group); EA8231 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Gemcitabine; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pembrolizumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (TPC chemotherapy) (Active Comparator): Patients receive TPC with carboplatin or cisplatin IV on day 1 and gemcitabine IV on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may alternately receive TPC with docetaxel IV on day 1 of each cycle or paclitaxel IV on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients additional undergo blood sample collection, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Other: Questionnaire Administration
- Arm II (pembrolizumab, sacituzumab govitecan) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and sacituzumab govitecan IV over 1-3 hours on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients additional undergo blood sample collection, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Other: Questionnaire Administration; Biological: Sacituzumab Govitecan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (TPC chemotherapy)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (TPC chemotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm I (TPC chemotherapy)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm I (TPC chemotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (TPC chemotherapy)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (pembrolizumab, sacituzumab govitecan)
Other: Questionnaire Administration — Ancillary studies
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU 132; IMMU-132; IMMU132; RS7 SN38; RS7-SN38; RS7SN38; Sacituzumab Govitecan-hziy; Trodelvy
  Arms: Arm II (pembrolizumab, sacituzumab govitecan)

SUMMARY:
This phase III trial compares the effectiveness of pembrolizumab and sacituzumab govitecan to standard of care in treating patients with urothelial cancer that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Sacituzumab govitecan is a monoclonal antibody, called sacituzumab, linked to a chemotherapy drug called govitecan. Sacituzumab attaches to TROP2 positive tumor cells in a targeted way and delivers govitecan to kill them. The usual treatment approach is treatment with chemotherapy such as cisplatin, carboplatin, gemcitabine, docetaxel or paclitaxel. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid and may kill tumor cells. Docetaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Giving pembrolizumab and sacituzumab govitecan may be more effective than usual care of carboplatin or cisplatin with gemcitabine, docetaxel or paclitaxel in treating patients with locally advanced or metastatic urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival (OS) between the therapy of physician choice (TPC) arm and the sacituzumab govitecan + pembrolizumab arm.

SECONDARY OBJECTIVES:

I. To compare the progression free survival (PFS) between the TPC arm and the sacituzumab govitecan + pembrolizumab arm.

II. To evaluate overall response rate (ORR) between the TPC arm and the sacituzumab govitecan + pembrolizumab arm.

III. To evaluate clinical benefit rate (complete response [CR]/partial response [PR] /stable disease [SD]) between the TPC arm and the sacituzumab govitecan + pembrolizumab arm.

IV. To evaluate duration of response (DoR) between the TPC arm and the sacituzumab govitecan + pembrolizumab arm.

V. To evaluate toxicity of the sacituzumab govitecan + pembrolizumab arm using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

EXPLORATORY HEALTH RELATED QUALITY OF LIFE (HRQOL) OBJECTIVES:

I. To compare HRQOL, as assessed by the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Bladder Symptom Index-18 (FBISI-18) summary score between patients on the TPC arm versus the sacituzumab govitecan + pembrolizumab arm at 6 months.

II. To compare HRQOL change from baseline, as assessed by the FBISI-18 summary score, for patients on the TPC arm versus the sacituzumab govitecan + pembrolizumab arm at baseline, 3, 6, and 12 months.

III. To compare the change in patient-reported fatigue from baseline and across 3, 6, and 12 months as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) summary score; change from baseline will be compared between patients on the TPC arm versus the sacituzumab govitecan + pembrolizumab arm.

IV. To compare quality-adjusted survival (overall survival x health utility score assessed by the European Quality of Life Five Dimension Five Level [EQ-5D-5L]) between patients on the TPC arm versus the sacituzumab govitecan + pembrolizumab arm.

V. To compare time to HRQOL deterioration in global HRQOL, as measured by the FBISI-18 disease-related physical symptom subscale (FBISI-18 disease-related symptoms (DRS) in the physical emotional domains [DRS-P]), between patients on the TPC arm versus the sacituzumab govitecan + pembrolizumab arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive TPC with carboplatin or cisplatin intravenously (IV) on day 1 and gemcitabine IV on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may alternately receive TPC with docetaxel IV on day 1 of each cycle or paclitaxel IV on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients additionally undergo blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

ARM B: Patients receive sacituzumab govitecan IV over 1-3 hours on days 1 and 8 and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 35 cycles or for 2 years of pembrolizumab in the absence of disease progression or unacceptable toxicity. Cycles of sacituzumab govitecan repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients additional undergo blood sample collection, and CT or MRI throughout the study.

After completion of study treatment, patients are followed up at 30 days then once a year for 5 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patient must have locally advanced (unresectable or not amenable to curative intent therapy) or metastatic urothelial cancer
* Patient must have histologically proven conventional urothelial carcinoma (UC) of any urinary tract origin [any histologic subtype except neuroendocrine (small or large cell)] are permitted so long as tumors include ≥ 1% urothelial histology). NOTE: Pure non-urothelial histology is excluded
* Patient must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Baseline imaging must be obtained ≤ 35 days prior to randomization
* Patient must have the following prior treatment. Patient must have had progression on or after the immediate prior therapy
* Patient must have had prior exposure to anti-PD(L)1 therapy [anti -PD(L)1 monotherapy or as a combination regimen in any disease/therapy setting for UC. Patients must have received at least 1 dose of anti-PD(L)1 therapy

  * NOTE: Anti-PD(L)1 therapy does not need to be the most recent therapy received prior to enrollment on this protocol
* Patient must not have had progression within 12 weeks of using anti-PD(l) 1 therapy
* Patient must have had ≥ 1 line of systemic therapy given in the advanced/metastatic disease setting. For tumors with FGFR3 + susceptible alteration (for FGFR inhibitor), patients must have received a prior FGFR inhibitor unless contraindicated per physician discretion
* Patient must have received prior enfortumab vedotin in any disease/therapy setting unless contraindicated per physician
* Patient must have had no prior exposure to sacituzumab govitecan or other TROP-2 directed therapies or antibody-drug conjugate that contains topo-isomerase I inhibitor, e.g. trastuzumab deruxtecan
* Patient must have Bellmunt score of 0-2. The Bellmunt score assesses a patient's risk and is calculated based upon ECOG PS, the hemogloblin level and presence of liver metastases
* Patient must not have any history of grade 3 or higher immune-related adverse events on prior anti-PD1/L1, except for endocrinopathies on adequate hormone therapy repletion and clinically insignificant laboratory abnormalities
* Patient must have recovered (i.e., ≤ grade 1) from clinically significant AEs due to previously administered systemic therapy agent, except for endocrinopathies on adequate hormone therapy repletion

  * NOTE: Patients with ≤ grade 2 neuropathy, any grade of alopecia, or any grade of non-clinically significant laboratory abnormality are exceptions to this criterion and are allowed in this trial.
  * Examples of non-clinically significant laboratory abnormalities include, but are not limited to:

    * Lymphopenia or monopenia
    * Lymphocytosis or monocytosis
    * Increase in amylase or lipase with no clinical correlation
    * Any other abnormal laboratory findings that have no clinical relevance per the treating investigators.
  * NOTE: If patient has undergone major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to randomization
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Patient must not nurse infants while on protocol treatment and for 4 months after the last dose of protocol treatment
* Patient must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. Patients of childbearing potential must continue contraceptive method(s) or abstain for 6 months after the last dose of protocol treatment. Patients with partners who could become pregnant should use effective contraception during therapy and for 3 months after the last dose of protocol treatment
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Absolute neutrophil count (ANC) ≥ 1,500/uL (obtained ≤ 14 days prior to randomization)
* Platelets ≥ 100,000/uL (obtained ≤ 14 days prior to randomization)
* Albumin ≥ 3 g/dL (obtained ≤ 14 days prior to randomization)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (obtained ≤ 14 days prior to randomization)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN or ≤ 5.0 x institutional ULN if known liver metastases (obtained ≤ 14 days prior to randomization)
* Creatinine clearance (CrCl) ≥ 30 mL/min (obtained ≤ 14 days prior to randomization) NOTE: CrCl is estimated using the Cockcroft-Gault formula (or can be measured by 24-hour urine collection if needed)
* Patient must not have a known genetic UGT1A1 deficiency (Gilbert's syndrome). Patients with variant type UGT1A1*28 allele may have increased levels of SN-38 metabolite (due to reduced SN-38 metabolism and clearance) and are at higher risk for severe adverse events when compared to wild-type.

  * NOTE: If a patient's UGT1A1 status is unknown, they are eligible to enroll (the study does not require this test as part of screening)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and considered cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and are not using steroids > 10 mg of prednisone (or equivalent) daily for brain metastases for at least 7 days prior to randomization
* Patients with a prior or concurrent malignancy that is not considered clinically significant and whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen (at the discretion of the treating physician) are eligible for this trial
* Patient must not be on systemic immunosuppressive medication, including steroids (if doses exceed the equivalent of prednisone 10 mg daily). Short courses of steroids, e.g. "burst", which are discontinued prior to randomization are acceptable. Patients on inhaled, intranasal, intra-articular and/or topical steroids are eligible
* Patient must be English or Spanish speaking to be eligible for the HRQOL component of the study.

  * NOTE: Sites cannot translate the associated HRQOL forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death due to any cause, assessed up to 5 years
  OS will be characterized with the method of Kaplan-Meier and will be compared between the two treatment arms using stratified log-rank test. The hazard ratio (HR) will be estimated, and a 95% confidence interval (CI) will be reported.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the earlier progression or death due to any cause, assessed up to 5 years
  PFS will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. PFS will be characterized with the method of Kaplan-Meier and will be compared between the two treatment arms using stratified log-rank test. The HR will be estimated, and a 95% CI will be reported.
Overall response rate (ORR) | Up to 5 years
  ORR will be assessed among patients who received at least one dose of protocol therapy using RECIST v 1.1 criteria. ORR will be defined as the number of patients with complete response (CR) and partial response (PR) divided by the number of treated patients. ORR will be calculated based on the definition by arm and will be reported with 95% CI.
Clinical benefit rate (CBR) | Up to 5 years
  CBR will be defined as CR, PR, or stable disease per RECIST v 1.1. CBR will be calculated based on the definition by arm and will be reported with 95% CI.
Duration of response (DOR) | From the first occurrence of a documented objective response to disease progression or death, whichever occurs first, assessed up to 5 years
  DOR will be assessed by RECIST v1.1. DOR will be characterized with the method of Kaplan-Meier and will be compared between the two treatment arms using stratified log-rank test. The HR will be estimated, and a 95% CI will be reported.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  AEs will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The percentage of patients with toxicities will be tabulated. The 90% CI for the true probability of observing toxicity of ≥ grade 4 on a given arm will be no wider than 12.3 %. The probability of observing ≥ 1 toxicity on a given arm with a true rate of 1% is 85.5%.

OTHER OUTCOMES:
Change in National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Bladder Symptom Index-18 (FBISI-18) summary score | At baseline and at 3, 6 and 12 months
  Change in patient reported FBISI-18 score will be compared between arms using a two-sample t-test. Assessment time will be considered as a continuous variable if there is a linear trend in quality of life (QOL) assessments over time or a set of dummy variables if a non-linear trend exists. Patient demographics and disease characteristics will be adjusted in the mixed effect model. A t-test will be performed to explore change of FBISI-18 summary score.
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) summary score | At baseline and at 3, 6 and 12 months
  Change in patient reported FACIT-F score will be compared between arms using a two-sample t-test. Mixed effect models will be constructed to estimate the time profile of FACIT-F in the two arms and to evaluate treatment-by-time interactions. Assessment time will be considered as a continuous variable if there is a linear trend in QOL assessments over time or a set of dummy variables if a non-linear trend exists. Patient demographics and disease characteristics will be adjusted in the mixed effect model.
Change in quality-adjusted survival (assessed by the European Quality of Life Five Dimension Five Level scale [EQ-5D-5L]). | At baseline and at 3, 6 and 12 months
  Change in patient reported EQ-5D-5L will be compared between the arms using a two-sample t-test. Quality-adjusted survival (assessed by the EQ-5D-5L), will be analyzed with quality-adjusted time without symptoms or toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (70):
- United States (70):
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Reading Hospital, West Reading, Pennsylvania
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm